CLINICAL TRIAL: NCT05312372
Title: A Phase 1/2, Open -Label, Multicenter Trial Investigating the Safety, Tolerability, Pharmacokinetics, and Preliminary Antineoplastic Activity of S095033 (MAT2A Inhibitor) in Combination With Paclitaxel in Participants With Advanced or Metastatic Esophageal Squamous Cell Carcinoma (ESCC)
Brief Title: S095033 in Combination With Paclitaxel as 2nd- or 3rd-line Treatment in Participants With Advanced or Metastatic ESCC
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Strategic development reasons
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL1-95033-002; 2022-000250-29 (EudraCT Number)
Record Dates: First submitted 2022-03-04; First posted 2022-04-05 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- S095033 in combination with paclitaxel (Experimental): Dose escalation - phase 1: S095033 will be administrated at dose of 100 mg,150 mg or 200 mg everyday during a 28-day cycle. The participants will also receive paclitaxel intravenously on D1, D8 and D15 last for 28 days.
  Dose expansion - phase 2: Participants with MTAP-deletion and those with MTAP-wild type tumors will be evaluated in separate and independent dose expansion subpopulations.S095033 will be administrated every day during a 28-day cycle at recommended phase 2 dose (RP2D). Paclitaxel given intravenously on D1, D8, and D15 during a 28-day cycle.
  Interventions: Drug: Combination (S095033 + paclitaxel)

INTERVENTIONS:
Drug: Combination (S095033 + paclitaxel) — Phase 1- dose escalation S095033 ; paclitaxel started at 80 mg/m²,(IV)
  Phase 2 - S095033 at RP2D; paclitaxel started at 80 mg/m²,(IV)

SUMMARY:
The purpose of this study is to determinate the safety profile, tolerability, pharmacokinetics, and preliminary antineoplastic activity of S095033 in combination with paclitaxel in participants with advanced or metastatic esophageal squamous cell carcinoma (ESCC)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant aged ≥ 18 years of age.
2. Estimated life expectancy ≥12 weeks.
3. Eastern Cooperative Oncology Group (ECOG) performance status < 2.
4. Women of childbearing potential (WOCBP) must use a highly effective method of birth control during study treatment until at least 6 months after the last dose of investigational medicinal product (IMP). In case of use of oral contraception, women should have been stable on the same contraceptive drug (i.e. same active principle) for at least 3 months prior to the first IMP administration.
5. Male participants with WOCBP partners must use a condom during the study and until at least 6 months after the last dose of IMP. In addition, contraception should be considered for their female partners. Contraceptive measures do not apply if the participant is sterile, vasectomized or sexually abstinent. Sperm donation will not be allowed during the study and for 6 months after the last dose of IMP.
6. Obtained informed consent (ICF) prior to any study-specific procedure.
7. Participants with histologically confirmed advanced or metastatic esophageal squamous cell carcinoma that has failed to respond to or has progressed after treatment with standard fluorouracil and platinum-based chemotherapy, or with an anti-PD1 or PD-L1 antibody and not previously treated with a taxane.
8. Participants who have received one or two prior lines of systemic therapy.
9. Documented progression on prior line of therapy.
10. Participants must have at least one measurable lesion, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 for solid tumors.
11. For participants with MTAP deletion, evidence of homozygous loss of MTAP in archival or fresh tumor tissue.
12. For participants with MTAP wild type, evidence of the presence of MTAP in archival or fresh tumor tissue.
13. Adequate hematological function based on the last assessment performed within 7 days prior to the first IMP administration.
14. Adequate coagulation function for all participants. For participants receiving anti- coagulant therapy (except platelet anti-aggregants), the adequate therapeutic levels of INR should be confirmed.
15. Adequate renal function based on the last assessment performed within 7 days prior to the first IMP administration.
16. Adequate hepatic function based on the last assessment performed within 7 days prior to the first IMP administration.
17. Serum albumin ≥ 3 g/dL.

Exclusion Criteria:

1. Non-ability to swallow oral medication.
2. Pregnant and lactating women.
3. WOCBP tested positive in a pregnancy test within 7 days prior to the first day of IMP administration.
4. Participation in another interventional study at the same time or within 2 weeks prior to the first IMP administration.
5. Participant already enrolled in the study (informed consent signed) and having received at least 1 dose of S095033 and/or paclitaxel.
6. Known prior severe hypersensitivity to investigational products or any component in their formulations.
7. Participants who have not recovered from toxicity of previous anticancer therapy, including Grade ≥ 1 non-hematologic toxicity, according to the National Cancer Institute Common Terminology Criteria for Adverse Event (NCI-CTCAE) version 5.0, prior to the first IMP administration.
8. Major surgery within 4 weeks prior to the first IMP administration or participants who have not recovered from side effects of the surgery.
9. Participants who do not have a biopsy (or sections of it) available or readily obtainable for central confirmation of MTAP status.
10. Have a history of Gilbert's syndrome.
11. History of gastrointestinal perforation and /or fistula or aorto-esophageal fistula within 6 months prior to randomization.
12. Apparent tumor invasion into organs located adjacent to the esophageal disease site (e.g. aorta or respiratory tract) at an increased risk of fistula in the study treatment assessed by investigator.
13. Have a degenerative retinal disease that could increase the risk for visual loss with S095033 or confound the interpretation of retinal changes in the course of S095033 treatment.
14. Severe or uncontrolled active acute or chronic infection.
15. Participants with a known clinically significant cardiovascular disease or condition.
16. Participants with thrombosis, or a history of deep vein thrombosis or pulmonary embolism, within 4 weeks prior to first IMP administration.
17. Symptoms suggesting central nervous system involvement, including symptomatic metastasis, for which treatment is required.
18. Participants who have received systemic anticancer treatment or radiotherapy less than 2 weeks before the first dose of S095033.
19. Any clinically significant medical condition (e.g. organ dysfunction) or laboratory abnormality likely to jeopardize the participant's safety or to interfere with the conduct of the study, in the investigator's opinion.
20. Any contraindication to the use of paclitaxel as per standard labelling and local guidance.
21. For prior and forbidden concomitant medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) associated with S095033 administration during the first cycle of treatment (Phase 1) | At the end of Cycle 1 (each cycle is 28 days)
  DLTs observed during a 28-day period
Adverse events (AEs) (Phase 1) | up to 28 days after the last IMP administration (for all AEs) or up to 4 years (for all SAE related to the research)
  Including adverse events (AEs) and serious adverse events (SAEs) according to NCI-CTCAE, version 5.0
Changes in laboratory assessments (hematology and blood biochemistry) (Phase 1) | Screening, Day1(D1) D8 D15 and D22 from Cycle 1 to Cycle 4 (each cycle is 28 days),D1 and D15 from Cycle 5 (each cycle is 28 days) up to 28 days after the last IMP administration
Changes in physical examination and in performance status (ECOG) (Phase 1) | Screening, D1 and D15 of Cycle 1, D1 for all the remaining cycles up to 28 days after the last IMP administration
Abnormalities in 12-lead ECG parameters (Phase 1) | Screening, D1 and D2 of Cycle 1, D1 for all the following cycles until withdrawal visit (within 5 days after the last IMP administration)
Changes in vital signs: SBP, DBP, respiratory rate and temperature (Phase 1) | Screening, D1 D8 D15 and D22 of Cycle 1, D1 for all the following cycles up to 28 days after the last IMP administration
Objective response per central review of antitumor activity (using Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1) (Phase 2) | Screening,and after the completion of every 2 cycles until disease progression

SECONDARY OUTCOMES:
The PK (pharmacokinetic) profile of S095033 and paclitaxel plasma concentration : Area under the plasma concentration-time curve (AUC) (Phase 1 and phase 2) | D1 D2 D8 D15 D28 of Cycle 1, D1 for the following cycles until the last IMP administration
The PK profile of S095033 and paclitaxel plasma concentration : Time to maximum concentration (Tmax) (Phase 1 and phase 2) | D1 D2 D8 D15 D28 of Cycle 1, D1 for the following cycles until the last IMP administration
The PK profile of S095033 and paclitaxel plasma concentration : Maximum plasma concentration (Cmax) (Phase 1 and phase 2) | D1 D2 D8 D15 D28 of Cycle 1, D1 for the following cycles until the last IMP administration
The PK profile of S095033 and paclitaxel plasma concentration : Trough concentation (Ctrough) (Phase 1 and phase 2) | : D1 D2 D8 D15 D28 of Cycle 1, D1 for the following cycles until the last IMP administration
The PK profile of S095033 and paclitaxel plasma concentration : Half time (t1/2) (Phase 1 and phase 2) | D1 D2 D8 D15 D28 of Cycle 1, D1 for the following cycles until the last IMP administration
The PK profile of S095033 and paclitaxel plasma concentration :apparent volume of distribution (Vd/F) (Phase 1 and phase 2) | D1 D2 D8 D15 D28 of Cycle 1, D1 for the following cycles until the last IMP administration
The PK profile of S095033 and paclitaxel plasma concentration :apparent clearance (CL/F) (Phase 1 and phase 2) | D1 D2 D8 D15 D28 of Cycle 1, D1 for the following cycles until the last IMP administration
Changes in plasma concentration of S-adenosylmethionine (SAM) and methionine (Phase 1 and phase 2) | D1 D2 D8 D15 D28 of Cycle 1, D1 for the following cycles until withdrawal visit (within 5 days after the last IMP administration)
Objective response per Investigator assessment of antitumor activity (using Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1) (Phase 1 and phase 2) | Screening, and after the completion of every 2 cycles until disease progression
Clinical Benefit (CB) (Phase 1 and phase 2) | Screening, and after the completion of every 2 cycles until disease progression
Duration of response (DOR) (Phase 1 and phase 2) | Screening, and after the completion of every 2 cycles until disease progression
Progression-free survival (PFS) (Phase 1 and phase 2) | Screening, and after the completion of every 2 cycles until disease progression
Overall survival (OS) (Phase 1 and phase 2) | Screening, and after the completion of every 2 cycles up to 6 months after the last IMP administration
Time To Response (TTR) (Phase 1 and phase 2) | Screening, and after the completion of every 2 cycles until the first occurrence of a complete response (CR) or partial response (PR), whichever occurs first
Adverse events (AEs) (Phase 2) | up to 28 days after the last IMP administration (for all AEs) or up to 4 years (for all SAE related to the research)
  Including adverse events (AEs) and serious adverse events (SAEs) according to NCI-CTCAE, version 5.0
DLT associated with S095033 administration during the first cycle of treatment (Phase 2) | At the end of Cycle1 (each cycle is 28 days)
  DLTs observed during a 28-day period
Changes in laboratory assessments (hematology and blood biochemistry ) (Phase 2) | Screening, D1, D8 D15 and D22 from Cycle 1 to Cycle 4 (each cycle is 28 days), D1 and D15 from Cycle 5 (each cycle is 28 days) up to 28 days after the last IMP administration
Changes in physical examination and in performance status (ECOG) (Phase 2) | Screening, D1 and D15 of Cycle 1, D1 for all the remaining cycles up to 28 days after the last IMP administration
Abnormalities in 12-lead ECG parameters (Phase 2) | Screening, D1 and D2 of Cycle 1, D1 for all the following cycles until withdrawal visit (within 5 days after the last IMP administration)
Changes in vital signs : SBP, DBP, respiratory rate and temperature (Phase 2) | Screening, D1 D8 D15 and D22 of Cycle 1, D1 for all the following cycles up to 28 days after the last IMP administration

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier.
  * with a first patient enrolled as of 1 January 2004 onwards.
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com/

REFERENCES:
- See also: Find Results on Servier Clinical Trial Data website — http://clinicaltrials.servier.com/